CLINICAL TRIAL: NCT00888160
Title: Timing of Orthopaedic Surgery in the Multiply-injured Patient: Development of a Protocol for Early Appropriate Care
Status: Completed | Type: Observational
Sponsor: MetroHealth Medical Center (Other)
Responsible Party: Principal Investigator, Heather A. Vallier, Professor of Orthopaedic Surgery, MetroHealth Medical Center
Other Study IDs: IRB06-00089
Record Dates: First submitted 2009-04-24; First posted 2009-04-27 (Estimated); Last update posted 2018-05-14 (Actual); Status verified 2017-03

CONDITIONS: Unstable Pelvic Ring Fracture; Unstable Acetabulum Fracture; Femur Fracture
MeSH Terms: conditions — Femoral Fractures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Early fixation of unstable fractures of the femur, pelvis, and acetabulum reduces some complication rates. However, in patients with multiple injuries, the optimal treatment of skeletal trauma may be affected by severe injury to the head, chest, or abdomen. The relationship between associated injury severity and the timing of definitive management of unstable fractures is not well-understood. The practice of "early total care," early definitive fracture management, has been criticized by some, who have suggested that additional hemorrhage with surgery may be associated with a deleterious systemic inflammatory response. The alternative extreme of "damage control orthopedics (DCO)" has been recently proposed as a means of providing provisional stability of major skeletal injury, generally through external fixation. It is speculated that DCO will diminish the potential for systemic compromise. However, the need for further (definitive) surgery on a delayed basis, and the potential additional complications and costs associated with this strategy are controversial. The investigators' goals are to define which injuries or parameters warrant delay of definitive orthopaedic care, and to determine what time interval for fracture fixation promotes optimal patient outcome. The investigators will assess the effects of fracture fixation on head injury, chest injury, abdominal injury, mortality, complications, patient outcomes, and costs.

ELIGIBILITY:
Inclusion Criteria:

* All patients at least 16 years of age treated at a major urban level 1 trauma center between the years 2000 and 2006, who had any of the following musculoskeletal injuries:

  * unstable pelvic ring fracture
  * unstable acetabulum fracture, or
  * femur fracture
* Patients will be included regardless of race or gender. Isolated fractures will be included

Exclusion Criteria:

* Low-energy pelvis and hip fractures will be excluded
* Patients younger than 16 years of age will be excluded

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients at least 16 years of age treated at a major urban level 1 trauma center between the years 2000 and 2006, who had any of the following musculoskeletal injuries: unstable pelvic ring fracture, unstable acetabulum fracture, or femur fracture.
Sampling Method: Probability Sample
Enrollment: 360 (Actual)
Dates: Start 2010-09 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2031-01

CONTACTS AND LOCATIONS:
Locations (1):
- MetroHealth Medical Center, Cleveland, Ohio, United States